CLINICAL TRIAL: NCT00566956
Title: Ultrasound-guided Hydrosalpinx Aspiration During Egg Collection Improves Pregnancy Outcome in In-vitro Fertilization: a Randomised Controlled Trial
Brief Title: Ultrasound-guided Hydrosalpinx Aspiration During Egg Collection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated because it is very difficult to recruit more patients.
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Responsible Party: Mr M Afnan, Assisted Conception Unit
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0288; CC/APM/DD/C2/05
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2007-11

CONDITIONS: Infertility
Keywords: Hydrosalpinx/IVF/Reproductive outcome.; Hydrosalpinx
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): For those assigned to Group 1, the hydrosalpinx will be aspirated after all the eggs have been collected, under GA. Under ultrasound-guidance, the aspiration (egg collection) needle will be inserted into the hydrosalpinx and suction applied until no more fluid is obtained. If there are bilateral hydrosalpinges, the process is repeated on the opposite side.
  Interventions: Procedure: Hydrosalpinx needle aspiration to arm 1
- 2 (No Intervention): Patients assigned to group 2 will not have the hydrosalpinx aspirated

INTERVENTIONS:
Procedure: Hydrosalpinx needle aspiration to arm 1 — For those assigned to Group I, the hydrosalpinx will be aspirated after all the eggs have been collected, under GA. Under ultrasound-guidance, the aspiration (egg collection) needle will be inserted into the hydrosalpinx and suction applied until no more fluid is obtained. If there are bilateral hydrosalpinges, the process is repeated on the opposite side. The hydrosalpinx fluid is discarded
  Arms: 1

SUMMARY:
· What we know: Hydrosalpinx and IVF About 40% of patients undergoing IVF have tubal disease and in 25%-30% of tubal disease patients there is fluid collection within the tube; hydrosalpinx. The amount of fluid in the hydrosalpinx is known to increase with ovarian stimulation (as in IVF) and often empties into the uterine cavity. Fluid from hydrosalpinges has been found to be detrimental to the growth and development of mouse embryos in vitro, and associated with reduced levels of endometrial integrins in vivo. This could be the explanation of the reduced pregnancy rates after IVF in patients with tubal disease and hydrosalpinx compared with those with tubal disease but no hydrosalpinx. This effect was evidence in both fresh and frozen embryo transfer cycles. Also there was a significant increase in miscarriage in association with hydrosalpinx.

The study aims to answer the question: does ultrasound-guided aspiration of ultrasound diagnosed hydrosalpinx at the time of egg collection improve the pregnancy rate in IVF?

DETAILED DESCRIPTION:
· What we do not know: Treatment of hydrosalpinx and IVF Several studies in the literature have suggested that the treatment of hydrosalpinx pre-IVF would improve the pregnancy rate to a level similar to tubal disease patients without hydrosalpinx. The treatment modalities explored were salpingectomy, salpingostomy, tubal occlusion and ultrasound-guided aspiration either one month before or at the time of egg collection. All studies reported to date have been retrospective and with poor control design. A prospective randomised controlled trial is needed. All modalities have been associated with a similar improvement in pregnancy rate, but the least invasive modality is ultrasound-guided aspiration at the time of oocyte collection. We propose to conduct a prospective randomised controlled trial to evaluate the effect of ultrasound-guided aspiration (versus no aspiration) of hydrosalpinx at the time of egg collection on the pregnancy rate in IVF.

ELIGIBILITY:
Inclusion Criteria:

* healthy women, ASA class 1 (normal healthy) or class 2 (with mild systemic disease);
* undergoing IVF or ICSI and reaching the stage of egg collection;
* with ultrasonically diagnosed hydrosalpinx and identifiable during the phase of ovarian stimulation;
* giving written informed consent.

Exclusion Criteria:

* patients not giving written informed consent;
* patients cancelled for poor ovarian response;
* ultrasonically diagnosed hydrosalpinx and identifiable for the first time at egg-collection

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 1999-10; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures were biochemical (urinary hCG test performed 14 days after embryo transfer) and clinical (presence of gestational sac by transvaginal ultrasound scan) pregnancy rates per randomised women. | 2-4 weeks

SECONDARY OUTCOMES:
Secondary outcome measures were implantation rate, first trimester miscarriages (any pregnancy loss before 12 weeks gestation) and pelvic infection. | 2-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Hammadieh, MD,MRCOG, Principal Investigator — Assisted Conception Unit
Locations (1):
- Assisted Conception Unit, Birmingham Women's Hospital, Birmingham University, Birmingham, United Kingdom

REFERENCES:
- [Result] Strandell A, Lindhard A, Waldenstrom U, Thorburn J, Janson PO, Hamberger L. Hydrosalpinx and IVF outcome: a prospective, randomized multicentre trial in Scandinavia on salpingectomy prior to IVF. Hum Reprod. 1999 Nov;14(11):2762-9. doi: 10.1093/humrep/14.11.2762. PMID 10548619
- [Derived] Hammadieh N, Coomarasamy A, Ola B, Papaioannou S, Afnan M, Sharif K. Ultrasound-guided hydrosalpinx aspiration during oocyte collection improves pregnancy outcome in IVF: a randomized controlled trial. Hum Reprod. 2008 May;23(5):1113-7. doi: 10.1093/humrep/den071. Epub 2008 Mar 13. PMID 18343810